CLINICAL TRIAL: NCT02680925
Title: The Influence of Lung Protective Ventilation During Pulmonary Lobectomy on Clinical Outcome in Pediatric Patients
Brief Title: Lung Protective Ventilation During Pulmonary Lobectomy in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, Associate professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: H1511-124-725
Record Dates: First submitted 2016-02-06; First posted 2016-02-12 (Estimated); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Pulmonary Complication

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional ventilation group (Placebo Comparator): Mechanical ventilation is maintained with tidal volume (TV) of 10 ml/kg without PEEP during two-lung ventilation and TV of 8 ml/kg without PEEP during one-lung ventilation. Alveolar recruitment is performed 3 times; after intubation, before one-lung ventilation and after lung resection.
  Interventions: Procedure: Conventional ventilation
- Lung protective ventilation group (Active Comparator): Mechanical ventilation is maintained with tidal volume (TV) of 6 ml/kg with PEEP 6 cmH2O during two-lung ventilation and TV of 4 ml/kg PEEP 6 cmH2O during one-lung ventilation. Alveolar recruitment is performed 3 times; after intubation, before one-lung ventilation and after lung resection.
  Interventions: Procedure: lung protective ventilation

INTERVENTIONS:
Procedure: lung protective ventilation — TV 4 ml/kg during one lung ventilation and 6 ml/kg during two-lung ventilation with PEEP of 6 cmH2O
  Arms: Lung protective ventilation group
Procedure: Conventional ventilation — TV 8 ml/kg during one lung ventilation and 10 ml/kg during two-lung ventilation without PEEP
  Arms: Conventional ventilation group

SUMMARY:
The investigator will evaluate the influence of lung protective ventilation on postoperative clinical outcome in pediatric patients. The hypothesis is that application of low tidal volume, intermittent alveolar recruitment and adequate positive end-expiratory pressure (PEEP) would be more beneficial than conventional ventilation in children.

ELIGIBILITY:
Inclusion Criteria:

* Children who are scheduled for lung lobectomy under general anesthesia
* ASA physical status I, II

Exclusion Criteria:

* History of airway or pulmonary interstitial disease
* Active URI
* Systemic inflammatory response disease
* cardiac disease

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 114 (Actual)
Dates: Start 2016-02; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
The number of patients with pulmonary complication | up to postoperative 7 days
  The number of patients with pulmonary complication including atelectasis, pulmonary infiltration, pulmonary edema, pulmonary infection, pleural effusion and pulmonary embolism

SECONDARY OUTCOMES:
The number of patients with desaturation | During surgery
  The number of patients with desaturation (SpO2 < 90%)
The number of patients with extrapulmonary complication | through study completion, an average of 1 year
Mean duration of mechanical ventilation | through study completion, an average of 1 year
Mean duration of ICU stay | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Tae Kim, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul national university hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee JH, Bae JI, Jang YE, Kim EH, Kim HS, Kim JT. Lung protective ventilation during pulmonary resection in children: a prospective, single-centre, randomised controlled trial. Br J Anaesth. 2019 May;122(5):692-701. doi: 10.1016/j.bja.2019.02.013. Epub 2019 Mar 8. PMID 30916035